CLINICAL TRIAL: NCT06845865
Title: Measurement of Intestinal Permeability in Intensive Care Patients With Single or Multiple Organ Failure
Acronym: BLUE-REA
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Centre Borelli UMR 9010 (Network)
Responsible Party: Sponsor
Other Study IDs: 2021PPRC02; 2023-A02005-40 (Other: Comité de protection des personnes Ouest IV)
Record Dates: First submitted 2025-02-11; First posted 2025-02-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: Multivisceral Failure Syndrome; Monovisceral Failure; Infection in ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with mono-organ failure: 20 < SAPS2 < 40
  Interventions: Dietary Supplement: enteric dyed solution
- patients with multi-visceral failure: 60 < SAPS2 < 80
  Interventions: Dietary Supplement: enteric dyed solution

INTERVENTIONS:
Dietary Supplement: enteric dyed solution — Oral administration of 0.5 mg/kg of body weight of food coloring dye

SUMMARY:
Multivisceral failure syndrome (MVFS) in humans is associated with a very high risk of mortality, ranging between 30 and 50%. This syndrome is associated with significant systemic inflammation and a high risk of bacteremia, the origin of which is not always identified. Among the possible causes of bacteremia, digestive translocation is the most probable but has not been formally proven to date. This translocation is made possible by the numerous cellular and metabolic alterations secondary to MVFS, which can lead to increased intestinal barrier permeability. Intestinal permeability is currently not systematically evaluated in clinical practice in humans.

This increased intestinal permeability, associated with the presence of inflammatory markers and a septic state, has been studied in several animal models ranging from the fruit fly (Drosophila) to the mouse. These studies have shown a high risk of mortality associated with increased intestinal permeability.

We propose to use this methodology in intensive care patients with at least one organ failure to investigate the link between increased intestinal permeability and survival chances.

ELIGIBILITY:
Inclusion Criteria:

Patient with single organ failure, secondary to sepsis, hospitalized in intensive care for a foreseeable duration of > 48 hours

* SAPS2 between 20 and 40 at the sixth hour after the diagnosis of organ failure.
* Consent from the patient or their trusted person.
* Affiliation to a social security system.
* Functional digestive tract and possible feeding (per os or via a nasogastric tube whose indication was determined independently of the study's needs).

Second group of patients with multi-organ failure:

* Multi-organ failure syndrome with at least 2 organ failures, secondary to sepsis.
* SAPS2 between 60 and 80 at the sixth hour after the diagnosis of organ failure.
* Consent from the patient or their trusted person.
* Affiliation to a social security system.
* Functional digestive tract and possible feeding (conscious patient able to swallow or with a nasogastric tube whose indication was determined independently of the study's needs).

Exclusion Criteria:

* Pregnant and breastfeeding women;
* Minors;
* Persons under administrative and judicial supervision;
* Absence of a functional digestive tract (patient unable to swallow and absence of a nasogastric tube, contraindication to enteral feeding);
* Patients with gastroparesis;
* Refusal of the patient or their trusted person;
* Patient with a SAPS2 at the sixth hour after the diagnosis of organ failure < 20 or between 40 and 60 or > 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hosptalized adults in ICU, France.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
intestinal failure and survival 90 days post inclusion | 2024-2027
  Evaluation of the impact of changes in permeability (classified into 3 categories: absent, moderately increased, and highly increased) on patient survival at day 90

SECONDARY OUTCOMES:
intestinal permeability as a function of organ failure | 2024-2027
  Comparison of average intestinal permeability between patients with a single organ failure versus multiple organ failures on day 1 in the blood (plasma)

CONTACTS AND LOCATIONS:
Overall Officials: Clément DUBOST, MD, PhD, Principal Investigator — National teaching army hospital BEGIN (Hôpital National d'Instruction des Armées BEGIN)
Locations (1):
- Hopital Bégin, Vincennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angarita SAK, Duarte S, Russell TA, Ruchala P, Elliott IA, Whitelegge JP, Zarrinpar A. Quantitative Measure of Intestinal Permeability Using Blue Food Coloring. J Surg Res. 2019 Jan;233:20-25. doi: 10.1016/j.jss.2018.07.005. Epub 2018 Jul 27. PMID 30502249
- [Background] Dambroise E, Monnier L, Ruisheng L, Aguilaniu H, Joly JS, Tricoire H, Rera M. Two phases of aging separated by the Smurf transition as a public path to death. Sci Rep. 2016 Mar 22;6:23523. doi: 10.1038/srep23523. PMID 27002861
- [Background] Doig CJ, Sutherland LR, Sandham JD, Fick GH, Verhoef M, Meddings JB. Increased intestinal permeability is associated with the development of multiple organ dysfunction syndrome in critically ill ICU patients. Am J Respir Crit Care Med. 1998 Aug;158(2):444-51. doi: 10.1164/ajrccm.158.2.9710092. PMID 9700119
- [Background] Gayat E, Cariou A, Deye N, Vieillard-Baron A, Jaber S, Damoisel C, Lu Q, Monnet X, Rennuit I, Azoulay E, Leone M, Oueslati H, Guidet B, Friedman D, Tesniere A, Sonneville R, Montravers P, Pili-Floury S, Lefrant JY, Duranteau J, Laterre PF, Brechot N, Chevreul K, Michel M, Cholley B, Legrand M, Launay JM, Vicaut E, Singer M, Resche-Rigon M, Mebazaa A. Determinants of long-term outcome in ICU survivors: results from the FROG-ICU study. Crit Care. 2018 Jan 18;22(1):8. doi: 10.1186/s13054-017-1922-8. PMID 29347987
- [Background] Harris CE, Griffiths RD, Freestone N, Billington D, Atherton ST, Macmillan RR. Intestinal permeability in the critically ill. Intensive Care Med. 1992;18(1):38-41. doi: 10.1007/BF01706424. PMID 1578045